CLINICAL TRIAL: NCT02583659
Title: The First-line Combined Chemotherapy for Advanced Gastric Cancer: A Prospective Observational Clinical Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianglin Yuan, Professor, Chief Physician, Huazhong University of Science and Technology
Other Study IDs: TJCC004
Record Dates: First submitted 2015-10-19; First posted 2015-10-22 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; First-line chemotherapy; Biomarker
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from peripheral blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Combined chemotherapy: AGC patients treated with first-line combined chemotherapy

SUMMARY:
This prospective cohort study aims to observe the efficacy and safety of the first-line combined chemotherapy for advanced gastric cancer(AGC) in Chinese population.

DETAILED DESCRIPTION:
1. Establish a clinical database for the advanced gastric cancer patients treated with first-line combined chemotherapy in Tongji hospital.

   1.1.Data including age, gender, smoking state, karnofsky performance score（KPS）, disease history, clinical stage, primary tumor site, metastasis site, surgery, first-line chemotherapy, therapy after failure of first-line treatment, radiotherapy, toxicity, survival time, the time of free of progress, response were collected.

   1.2.The peripheral blood samples were collected for further biomarker reserch.
2. Kaplan-Meier and Cox model will be used to analyze the overall survival(OS) and progression-free survival(PFS) of advanced gastric cancer.
3. Extract Deoxyribonucleic acid（DNA） from the the peripheral blood and research biomarkers related to the first-line combined chemotherapy for AGC.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathology or cytopathology proven gastric cancer or gastroesophageal adenocarcinoma;
2. Unresectable locally advanced, or recurrent, or metastasis disease；
3. Chemotherapy-naive or disease progress at least 6 months after adjuvant chemotherapy completed.
4. Life expectancy of at least 3 months;
5. ECOG score 0-2;
6. Voluntarily signed the informed consent.

Exclusion criteria:

1. Previously treated with first-line chemotherapy;
2. First-line chemotherapy with single drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histopathology or cytopathology confirmed unresectable locally advanced, or recurrent, or metastatic chemotheapy-naive gastric cancer and gastroesophageal adenocarcinoma patients
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-06 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) . overall survival Overall survival(OS) | From date of enrollment until the date of death from any cause, assessed up to 60 months

SECONDARY OUTCOMES:
Progression-free survival(PFS) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Objective response rate(ORR) | The sum of complete remission (CR) rate and partial remission (PR) rate. Response will be measured through first-line treatment completion, up to 1 year
Disease control rate(DCR) | The sum of CR rate, PR rate and stable disease(SD) rate. Response will be measured through first-line treatment completion, up to 1 year
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Through first-line treatment completion,up to 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Xianglin Yuan, MD,PHD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China